CLINICAL TRIAL: NCT05536531
Title: Role of Neuromuscular Electrical Stimulation to Prevent Respiratory Muscle Weakness in Critically Ill Patients and Its Association to Changes in Myokines Profile. a Randomized Clinical Trial.
Brief Title: NMES Role to Prevent Respiratory Muscle Weakness in Critically Ill Patients and Its Association to Changes in Myokines.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 52-c50; ID 210602003 (Other Grant/Funding Number: Health Science Department Grant IV-2020)
Record Dates: First submitted 2022-07-20; First posted 2022-09-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-07

CONDITIONS: Muscle Weakness or Atrophy; Mechanical Ventilation Complication; Electrical Stimulations
Keywords: Neuromuscular electrical stimulation; Critical care
MeSH Terms: conditions — Muscle Weakness; Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Analysis of respiratory function (diaphragm) derived from Twitch maneuver and echography (posterior images analysis) will be performed blind to arm assignment. Given sedation, patients will be also be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES group (Experimental): NMES will be implemented simultaneously on quadriceps femoris muscles of both lower limbs using an electrical stimulator (TRAINFES 6 ADVANCED, Biomedical devices Spa, Santiago, Chile). Four rubber surface electrodes will be placed over motor points. However, since the electrodes will cover big proportion of muscle surface, anatomical distribution of the belly muscle plus visible contraction of it will be considered for correct setting. The stimulation will be delivered by biphasic current, symmetric (compensated) impulses of 45-50 Hz frequency, 400 μsec pulse duration. With a stimulus duration of 25 minutes, and an on-off programming of 5 seconds on (including 0.8 second rise time, 3.4 seconds of plateau and 0.8 second of fall time) and 5 seconds off, at current intensities able to cause maximal visible contractions. The session duration will be 30 minutes and will be applied twice a day.
  Interventions: Device: Neuromuscular electrical stimulation (NMES)
- Control (No Intervention): Sham NMES will not be provided. Standard care won´t be altered and passive mobilization will be performed according to routine ICU procedures.

INTERVENTIONS:
Device: Neuromuscular electrical stimulation (NMES) — Electrical stimulator (Electrostimulator TRAINFES 6 ADVANCED, Biomedical devices Spa, Santiago, Chile.) to administer NMES
  Other Names: Standard Care
  Arms: NMES group

SUMMARY:
Particularly, muscle respiratory wasting will occur early (18 to 69 hours) in up to 60% of patients with mechanical ventilation (MV), leading rapidly to diaphragmatic weakness, which is associated with prolonged MV use, longer ICU and hospital stay, and higher mortality risk. Sepsis and muscle inactivity, derived from sedation and MV use, are key driver mechanisms for developing these consequences, which can be avoided through early physical activation. However, exercise is limited at the early stages of care, where sedation and MV are needed, delaying muscle activation. Neuromuscular electrical stimulation (NMES) represents an alternative to achieve early muscle contraction in non-cooperative patients, being able to prevent local muscle wasting and, according to some reports, has the potential to shorten the time on MV, suggesting a systemic effect through myokines, a diverse range of cytokines and chemokines secreted by myocytes during muscle contraction. However, no studies have evaluated whether NMES applied to peripheral muscles can exert distant muscle effects over the diaphragm, ameliorating its weakness and if this protective profile is associated with myokine's change in ICU patients. This proposal comprises a randomized controlled study of NMES applied twice daily, for three days, compared to standard care (no NMES). Thirty-two patients will be recruited in the first 48 hours after MV and randomly assigned to the control group or NMES group (16 subjects each). Muscle characterization of quadriceps and diaphragm will be performed at baseline (Day 1, before the first NMES session) and after the last NMES session (morning of day 4). Myokine measurements [IL-1, IL-6, IL-15, Brain-Derived Neurotrophic Factor (BDNF), Myostatin and Decorin], through blood serum obtained from peripheric blood samples, will be performed just before starting NMES (T0) at the end of the session (T0.5), and 2 and 6 hours later (T2 and T6). These myokine curves will be repeated on days 1 and 3 at the first NMES session of the day. The Control group will be assessed in the same way and timing, except that blood samples will be at T0 and T6. Additionally, functional outcomes such as MV time and ICU length of stay will be registered for all patients at ICU discharge. Standard care won´t be altered.

DETAILED DESCRIPTION:
Critically ill patients hospitalized at Intensive Care Units (ICU) are characterized by an accelerated muscle wasting, which leads to general muscle weakness and loss of physical functions even after discharge. Particularly, muscle respiratory wasting will occur early (18 to 69 hours) in up to 60% of patients with mechanical ventilation (MV), leading rapidly to diaphragmatic weakness, which is associated with prolonged MV use, longer ICU and hospital stay and higher mortality risk. Sepsis and muscle inactivity, derived from sedation and MV use, are key driver mechanisms to developing these negative consequences, which can be avoided through early physical activation. However, exercise is limited at early stages of care, where sedation and MV are needed, delaying muscle activation and favoring a vicious circle.

Neuromuscular electrical stimulation (NMES) represents an alternative to achieve early muscle contraction in non-cooperative patients, being able to prevent local muscle wasting and, according to some reports, has the potential to shorten the time on MV, suggesting a systemic effect through myokines, a diverse range of cytokines and chemokines secreted by myocytes during muscle contraction. These factors modulate the function and metabolism of distant organs and can promote muscle cell proliferation and growth in order to maintain muscle structure and function. However, no studies have evaluated whether NMES applied to peripheral muscles can exert distant muscle effects over the diaphragm, ameliorating its weakness, and if this protective profile is associated to myokine's change in critically ill patients.

We hypothesize that in mechanical ventilated ICU patients NMES contributes to prevent respiratory muscle weakness when initiated at an early phase of their critical illness, and this effect is associated to acute changes in myokine profile, being able to facilitate discontinuation of MV and decrease ICU length of stay.

This proposal comprises a randomized controlled study of NMES applied twice a day, for 3 days, in comparison to standard care (no NMES). Thirty-two patients will be recruited in the first 48 hours after connection to MV, and randomly assigned to either control group or stimulated group (16 subjects for each group). Muscle characterization of quadriceps and diaphragm (Structural ultrasonography evaluation of muscle thickness and tracheal twitch pressure assessment, derived from magnetic stimulation of phrenic nerve, for diaphragmatic strength) will be performed at baseline (Day 1, prior to the first NMES session) and after the last NMES session (morning of day 4). Myokine measurements (IL-1, IL-6, IL-15, BDNF, Myostatin and Decorin), through blood serum obtained from peripheric blood samples, will be performed at baseline 1 hour before NMES (T-1), just before starting NMES (T0), at the end of NMES session (T0.5), and 2 and 6 hours later (T2 and T6). This myokine curves will be repeated on days 1 and 3 at the first NMES session of the day. Control group will be assessed in the same way and timing, with the exception that blood samples will be performed at T0 and T6 of days 1 and 3. Additionally, functional outcomes such as MV time and ICU length of stay will be registered for all patients at ICU discharge. Standard care won´t be altered, performing passive mobilization according to ICU procedures in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutively admission to Christus ICU between March 2021 and December 2021.
2. Connected to invasive MV within the previous 24-48 hours
3. Deep sedation [non-cooperative state; Sedation-Agitation Scale (SAS) 1 or 2].
4. ICU-acquired weakness risk (One of the following risk factors: the need for invasive MV, sepsis, hyperglycemia, APACHE II admission score >13 pts, use of corticosteroids, and/or muscle inactivity due to deep sedation).
5. Written informed consent provided by patient/surrogate

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Obesity (Body Mass Index >35 kg/m2)
4. Pre-existing Neuromuscular diseases (e.g., myasthenia Gravis, Guillain-Barré disease)
5. Diseases with systemic vascular involvement such as systemic lupus erythematosus.
6. Use of neuromuscular blockers
7. Technical obstacles to the implementation of NMES such as bone fractures or skin lesions (e.g., burns)
8. End-stage malignancy
9. Presence of cardiac pacemakers
10. Diagnosis of brain death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Tracheal twitch pressure (centimeters of water) | Change from begining (Day one) and at the end (Day three)
  Sub Maximal diaphragmatic strength measured trough tracheal twitch pressure derived from magnetic stimulation of phrenic nerve.
Change in Diaphragmatic thickness fraction (centimeter percentage change) | Change from begining (Day one) and at the end (Day three)
  Diaphragmatic function derived from ultrasonography measurement of diaphragmatic muscle thickness between inspiration and expiration (during twitch manoeuvre)

SECONDARY OUTCOMES:
IL-1 myokine | through Study, at begining (Day one) and at the end (Day three). Before and after intervención
  IL-1 Measured in peripheral blood samples (pg/dL)
IL-6 myokine | through Study, at begining (Day one) and at the end (Day three). Before and after intervención
  IL-6 Measured in peripheral blood samples (pg/dL)
Decorin myokine | through Study, at begining (Day one) and at the end (Day three). Before and after intervención
  Decorin Measured in peripheral blood samples (pg/dL)
Myostatin myokine | through Study, at begining (Day one) and at the end (Day three). Before and after intervención
  Myostatin Measured in peripheral blood samples (pg/dL)
IL-15 myokine | through Study, at begining (Day one) and at the end (Day three). Before and after intervención
  IL-15 Measured in peripheral blood samples (pg/dL)
Brain derived neurotrophic Factor (BDNF) myokine | through Study, at begining (Day one) and at the end (Day three). Before and after intervención
  BDNF Measured in peripheral blood samples (pg/dL)
Change in Diaphragmatic muscle structure (cemtimeters) | Change from begining (Day one) and at the end (Day three)
  Diaphragmatic thickness measured with ultrasonography (Centimeters)
Change in peripheral muscle structure (centimeters) | Change from begining (Day one) and at the end (Day three)
  Muscle layer thickness of vastus intermedius and rectus femoris of the quadriceps, measured with ultrasonography (Centimeters)
Functional outcomes | through Study completion, an average of 1 month as maximum during follow up
  Mechanical Ventilation time (Hours)
Functional outcomes | through Study completion, an average of 2 month as maximum during follow up
  ICU length of stay (Days)

CONTACTS AND LOCATIONS:
Overall Officials: Yorschua Jalil, PT, MSc, Principal Investigator — Facultad de Medicina, Pontificia Universidad Católica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Dres M, Dube BP, Mayaux J, Delemazure J, Reuter D, Brochard L, Similowski T, Demoule A. Coexistence and Impact of Limb Muscle and Diaphragm Weakness at Time of Liberation from Mechanical Ventilation in Medical Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Jan 1;195(1):57-66. doi: 10.1164/rccm.201602-0367OC. PMID 27310484
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Dirks ML, Hansen D, Van Assche A, Dendale P, Van Loon LJ. Neuromuscular electrical stimulation prevents muscle wasting in critically ill comatose patients. Clin Sci (Lond). 2015 Mar;128(6):357-65. doi: 10.1042/CS20140447. PMID 25296344
- [Background] Truong AD, Kho ME, Brower RG, Feldman DR, Colantuoni E, Needham DM. Effects of neuromuscular electrical stimulation on cytokines in peripheral blood for healthy participants: a prospective, single-blinded Study. Clin Physiol Funct Imaging. 2017 May;37(3):255-262. doi: 10.1111/cpf.12290. Epub 2015 Oct 16. PMID 26475418
- [Background] Routsi C, Gerovasili V, Vasileiadis I, Karatzanos E, Pitsolis T, Tripodaki E, Markaki V, Zervakis D, Nanas S. Electrical muscle stimulation prevents critical illness polyneuromyopathy: a randomized parallel intervention trial. Crit Care. 2010;14(2):R74. doi: 10.1186/cc8987. Epub 2010 Apr 28. PMID 20426834